CLINICAL TRIAL: NCT02716662
Title: Safety of Caprylic Triglycerides in ALS: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Dr. Dale J. Lange, MD, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1307014081
Record Dates: First submitted 2016-01-06; First posted 2016-03-23 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: ALS
MeSH Terms: interventions — caprylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): Axona
  Interventions: Dietary Supplement: Axona

INTERVENTIONS:
Dietary Supplement: Axona — medical powder, supplement food
  Other Names: AC1204

SUMMARY:
The purpose of this study is to determine if AC-1204 is safe and tolerated in subjects with ALS. The reason why the investigator wants to use AC-1204 in patients with ALS is to determine if, by taking AC-1204, the body will make substances called ketone bodies. Further, if AC-1204 is well tolerated, the investigators want to change the amount the participant takes, to determine if the amount of ketone bodies in the blood increase in accordance with increases in the amount of AC-1204 the participant takes. The investigators want to do this study because when the investigators gave AC-1204 to mice with ALS, findings suggest the disease course is altered for the better and that the cause of this change is due to the presence of ketones in the blood. If AC-1204 can be proven to be safe and able to cause ketones to increase in the blood, the investigators will likely do subsequent studies to determine if the presence of ketone bodies will slow or stop the progression of the disease. However, this study is not designed to determine if AC-1204 will stop or slow the progression of ALS. It is designed to only determine if patients with ALS can tolerate AC-1204, if ketone bodies are produced and if the amount of ketone bodies produced increases with increasing dose.

ELIGIBILITY:
Inclusion Criteria:

* Familial or sporadic ALS diagnosed as probable, laboratory-supported probable or definite according to the World Federation of Neurology El Escorial criteria,
* Age 18 or older,
* Capable of providing informed consent and complying with trial procedures,
* Appel ALS score less than 100,
* Able to stand on a scale with assistance,
* Willing to chart food intake during the 12 week study,
* Patients either not taking Riluzole (Rilutek) or on a stable dose for 30 days or more,
* Not taking Coenzyme Q10 or on a stable dose and brand for 30 days,
* Absence of exclusion criteria.

Exclusion Criteria:

* Forced vital capacity <40% of predicted,
* Dependence on mechanical ventilation for more than 12 hours per day,
* Exposure to any experimental agent within 30 days of entry or at any time during the trial,
* Women who are breastfeeding, who are pregnant or are planning to become pregnant,
* Women of childbearing potential not practicing a medically accepted form of contraception,
* Enrollment in another research study within 30 days of or during this trial,
* Mini-Mental State Exam (MMSE) score <20,
* Patients with symptomatic cardiac disease or hypercholesterolemia,
* Patients with myocardial infarction within 6 months of this trial,
* Renal dysfunction defined as BUN and creatinine >2xULN,
* Known mitochondrial disease,
* BMI<18.5,
* Prior use of a 4:1 ketogenic diet or Atkins diet within 1 month of this trial,
* Impaired liver function, defined as AST or ALT of 3xULN,
* Patients who have a pacemaker or other internal electronic medical device,
* Known allergy or hypersensitivity to milk or soy products.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Ketone levels | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States